CLINICAL TRIAL: NCT01732796
Title: A Phase III, Randomized, Partially Double-Blind and Placebo-Controlled Study of BI 207127 in Combination With Faldaprevir and Ribavirin in Treatment-Naive Patients With Chronic Genotype 1 HCV Infection
Brief Title: IFN-free Combination Therapy in HCV-infected Patients Treatment-naive:HCVerso1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1241.20; 2012-003533-41 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-11-06; First posted 2012-11-26 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; faldaprevir; deleobuvir

ARMS (3):
- Allocated 24 weeks BI 207127 + BI 201335 (Experimental): 24 weeks of BI 207127 and BI 201335 in combination with Ribavirin
  Interventions: Drug: Ribavirin (RBV); Drug: BI 201335 (Faldaprevir); Drug: BI 207127
- Randomized 16 weeks BI 7127+BI1335 + RBV (Experimental): 16 weeks of BI 207127 and QD BI 201335 RBV, followed by additional 8 weeks of placebo BI 207127+ placebo BI 201335 in combination with placebo RBV
  Interventions: Drug: BI 201335 (Faldaprevir); Drug: Ribavirin (RBV); Drug: BI 207127
- Randomized 24weeks BI 7127+ BI1335 + RBV (Experimental): 24 weeks of BI 207127and BI 201335 in combination with RBV
  Interventions: Drug: Ribavirin (RBV); Drug: BI 207127; Drug: Faldaprevir (BI 201335)

INTERVENTIONS:
Drug: Ribavirin (RBV) — 24 weeks of active RBV
  Arms: Allocated 24 weeks BI 207127 + BI 201335
Drug: BI 201335 (Faldaprevir) — 16 weeks of BI 201335 followed by 8 weeks placebo to BI 201335
  Arms: Randomized 16 weeks BI 7127+BI1335 + RBV
Drug: Ribavirin (RBV) — 24 weeks of active RBV
  Arms: Randomized 24weeks BI 7127+ BI1335 + RBV
Drug: BI 207127 — 24 weeks of BI 207127
  Arms: Randomized 24weeks BI 7127+ BI1335 + RBV
Drug: BI 201335 (Faldaprevir) — 24 weeks of BI 201335
  Arms: Allocated 24 weeks BI 207127 + BI 201335
Drug: Ribavirin (RBV) — 16 weeks of Ribavirin followed by 8 weeks of placebo to Ribavirin
  Arms: Randomized 16 weeks BI 7127+BI1335 + RBV
Drug: BI 207127 — 16 weeks BI 207127 followed by 8 weeks placebo to BI 207127
  Arms: Randomized 16 weeks BI 7127+BI1335 + RBV
Drug: Faldaprevir (BI 201335) — 24 weeks of 201335
  Arms: Randomized 24weeks BI 7127+ BI1335 + RBV
Drug: BI 207127 — 24 weeks of BI 207127
  Arms: Allocated 24 weeks BI 207127 + BI 201335

SUMMARY:
The aim of the study is to confirm efficacy of treatment for 16 and 24 weeks in chronically infected HCV GT1b treatment naïve patients, including patients with compensated cirrhosis.

ELIGIBILITY:
Inclusion criteria:

* Chronic hepatitis C infection, diagnosed by positive HCV Ab or detectable HCV RNA at screening in addition to at least one of the following:

  1. positive HCV RNA or HCV antibodies at least 6 months prior to screening, or
  2. liver biopsy typical of chronic hepatitis C , or
  3. history of elevated ALT at least 6 months prior to screening.
* HCV infection of sub-GT1b confirmed by genotypic testing at screening
* Treatment naïve defined as:

  1. no prior treatment with any interferon, pegylated interferon, and /or ribavirin and
  2. no prior treatment with at least one dose of any other licensed or investigational antiviral agent for acute or chronic hepatitis C infection
* Plasma HCV RNA > or = 1,000 IU/mL at screening
* Liver biopsy within three years or fibroscan within six months prior to randomization. Patients with compensated liver cirrhosis (score Child-Pugh A) could also be included.
* Age 18 to 75 years
* Female patients with a negative urine pregnancy test (dipstick) at Visit 2 prior to randomization

  1. with documented hysterectomy, or
  2. who have had both ovaries removed, or
  3. with documented tubal ligation, or
  4. who are post-menopausal with last menstrual period at least 12 months prior to screening, or
  5. of childbearing potential with a negative serum pregnancy test at screening and a negative urine pregnancy test on Day 1 (Visit 2), that agree to use two non-hormonal methods of birth control from the date of screening until months after the last dose of ribavirin. They must not breast-feed at any time from the date of screening until 7 months after the last dose of ribavirin. Medically accepted methods of contraception for females in this trial are diaphragm with spermicide substance, intrauterine devices, cervical caps and condoms.

OR:

Male patients

1. who are documented to be sterile, or
2. who consistently and correctly use a condom while their female partners (if of child-bearing potential) agree to use one of the appropriate medically accepted methods of birth control from the date of screening until 7 months after the last dose of ribavirin, and
3. without pregnant female partners. It is in the responsibility of the male patient to ensure that his partner (or partners) is not pregnant prior to enrolment into the study or becomes pregnant during the treatment and follow-up phase. Female partners of childbearing potential must perform monthly pregnancy tests from the date of screening until 7 months after the last dose of ribavirin (tests will be provided by the sponsor).

Exclusion criteria:

* HCV infection of mixed genotype (1/2, 1/3, and 1/4) diagnosed by genotypic testing at screening.
* HCV subtype 1a, mixed 1a/1b or GT1 undefined
* Evidence of liver disease mainly due to causes other than chronic HCV infection such as autoimmune hepatitis, primary biliary cirrhosis, hemochromatosis or Wilson's disease
* HIV-1 or HIV-2 infection
* Hepatitis B virus (HBV) infection based on presence of HBs-Ag
* Evidence of decompensated liver disease, or history of decompensated liver disease, defined as history of ascites, hepatic encephalopathy, or bleeding esophageal varices,
* International Normalized Ratio (INR) > or =1.7
* Serum albumin < 3.3 g/dL
* Serum total bilirubin >2.0 times the upper limit of normal (ULN) with direct/indirect ratio >1, unless history of Gilbert's disease
* Active or suspected malignancy or history of malignancy within the last 5 years (with the exception of appropriately treated basal cell carcinoma of the skin or in situ carcinoma of the uterine cervix)
* Patients with ongoing or historical photosensitivity or recurrent rash

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2012-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (101):
- United States (24):
  - 1241.20.00026 Boehringer Ingelheim Investigational Site, Dothan, Alabama
  - 1241.20.00033 Boehringer Ingelheim Investigational Site, Chula Vista, California
  - 1241.20.00006 Boehringer Ingelheim Investigational Site, La Mesa, California
  - 1241.20.00003 Boehringer Ingelheim Investigational Site, Oceanside, California
  - 1241.20.00008 Boehringer Ingelheim Investigational Site, Poway, California
  - 1241.20.00015 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1241.20.00014 Boehringer Ingelheim Investigational Site, Ft. Pierce, Florida
  - 1241.20.00004 Boehringer Ingelheim Investigational Site, Maitland, Florida
  - 1241.20.00010 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 1241.20.00001 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 1241.20.00018 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1241.20.00002 Boehringer Ingelheim Investigational Site, Chevy Chase, Maryland
  - 1241.20.00032 Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - 1241.20.00009 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1241.20.00016 Boehringer Ingelheim Investigational Site, New York, New York
  - 1241.20.00031 Boehringer Ingelheim Investigational Site, New York, New York
  - 1241.20.00019 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1241.20.00024 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 1241.20.00013 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1241.20.00005 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1241.20.00017 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1241.20.00012 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1241.20.00022 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1241.20.00020 Boehringer Ingelheim Investigational Site, Richmond, Virginia
- 1241.20.43003 Boehringer Ingelheim Investigational Site, Graz, Austria
- Canada (8):
  - 1241.20.01001 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1241.20.01008 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1241.20.01010 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1241.20.01003 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1241.20.01006 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1241.20.01002 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1241.20.01005 Boehringer Ingelheim Investigational Site, Whitby, Ontario
  - 1241.20.01007 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- France (9):
  - 1241.20.33003 Boehringer Ingelheim Investigational Site, Clermont-Ferrand
  - 1241.20.33004 Boehringer Ingelheim Investigational Site, Lyon
  - 1241.20.33006 Boehringer Ingelheim Investigational Site, Marseille
  - 1241.20.33001 Boehringer Ingelheim Investigational Site, Montpellier
  - 1241.20.33005 Boehringer Ingelheim Investigational Site, Nice
  - 1241.20.33007 Boehringer Ingelheim Investigational Site, Paris
  - 1241.20.33002 Boehringer Ingelheim Investigational Site, Pessac
  - 1241.20.33009 Boehringer Ingelheim Investigational Site, Rennes
  - 1241.20.33008 Boehringer Ingelheim Investigational Site, Vandœuvre-lès-Nancy
- Germany (14):
  - 1241.20.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 1241.20.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 1241.20.49012 Boehringer Ingelheim Investigational Site, Bonn
  - 1241.20.49013 Boehringer Ingelheim Investigational Site, Cologne
  - 1241.20.49001 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1241.20.49014 Boehringer Ingelheim Investigational Site, Hamburg
  - 1241.20.49009 Boehringer Ingelheim Investigational Site, Herne
  - 1241.20.49008 Boehringer Ingelheim Investigational Site, Kiel
  - 1241.20.49011 Boehringer Ingelheim Investigational Site, Leipzig
  - 1241.20.49006 Boehringer Ingelheim Investigational Site, Magdeburg
  - 1241.20.49003 Boehringer Ingelheim Investigational Site, München
  - 1241.20.49010 Boehringer Ingelheim Investigational Site, Oberhausen
  - 1241.20.49005 Boehringer Ingelheim Investigational Site, Ulm
  - 1241.20.49007 Boehringer Ingelheim Investigational Site, Würzburg
- Hungary (2):
  - 1241.20.36001 Boehringer Ingelheim Investigational Site, Budapest
  - 1241.20.36002 Boehringer Ingelheim Investigational Site, Kaposvár
- Ireland (3):
  - 1241.20.35301 Boehringer Ingelheim Investigational Site, Dublin
  - 1241.20.35302 Boehringer Ingelheim Investigational Site, Dublin
  - 1241.20.35303 Boehringer Ingelheim Investigational Site, Dublin
- Italy (8):
  - 1241.20.39007 Boehringer Ingelheim Investigational Site, Ancona
  - 1241.20.39003 Boehringer Ingelheim Investigational Site, Brescia
  - 1241.20.39002 Boehringer Ingelheim Investigational Site, Milan
  - 1241.20.39008 Boehringer Ingelheim Investigational Site, Milan
  - 1241.20.39006 Boehringer Ingelheim Investigational Site, Napoli
  - 1241.20.39005 Boehringer Ingelheim Investigational Site, Pavia
  - 1241.20.39001 Boehringer Ingelheim Investigational Site, Torino
  - 1241.20.39004 Boehringer Ingelheim Investigational Site, Torino
- Netherlands (5):
  - 1241.20.31001 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1241.20.31003 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1241.20.31004 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1241.20.31005 Boehringer Ingelheim Investigational Site, Groningen
  - 1241.20.31006 Boehringer Ingelheim Investigational Site, The Hague
- Portugal (5):
  - 1241.20.35103 Boehringer Ingelheim Investigational Site, Aveiro
  - 1241.20.35104 Boehringer Ingelheim Investigational Site, Coimbra
  - 1241.20.35101 Boehringer Ingelheim Investigational Site, Lisbon
  - 1241.20.35102 Boehringer Ingelheim Investigational Site, Porto
  - 1241.20.35105 Boehringer Ingelheim Investigational Site, Vila Real
- Romania (3):
  - 1241.20.40001 Boehringer Ingelheim Investigational Site, Bucharest
  - 1241.20.40002 Boehringer Ingelheim Investigational Site, Bucharest
  - 1241.20.40003 Boehringer Ingelheim Investigational Site, Bucharest
- Russia (4):
  - 1241.20.70002 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 1241.20.70001 Boehringer Ingelheim Investigational Site, Moscow
  - 1241.20.70004 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1241.20.70005 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Spain (8):
  - 1241.20.34007 Boehringer Ingelheim Investigational Site, A Coruña
  - 1241.20.34004 Boehringer Ingelheim Investigational Site, Alicante
  - 1241.20.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1241.20.34005 Boehringer Ingelheim Investigational Site, Barcelona
  - 1241.20.34003 Boehringer Ingelheim Investigational Site, Madrid
  - 1241.20.34001 Boehringer Ingelheim Investigational Site, Majadahonda, Madrid
  - 1241.20.34008 Boehringer Ingelheim Investigational Site, Santander
  - 1241.20.34006 Boehringer Ingelheim Investigational Site, Valencia
- United Kingdom (7):
  - 1241.20.44005 Boehringer Ingelheim Investigational Site, Bristol
  - 1241.20.44007 Boehringer Ingelheim Investigational Site, Liverpool
  - 1241.20.44001 Boehringer Ingelheim Investigational Site, London
  - 1241.20.44002 Boehringer Ingelheim Investigational Site, London
  - 1241.20.44006 Boehringer Ingelheim Investigational Site, London
  - 1241.20.44004 Boehringer Ingelheim Investigational Site, Nottingham
  - 1241.20.44003 Boehringer Ingelheim Investigational Site, Southampton

REFERENCES:
- [Derived] Sarrazin C, Castelli F, Andreone P, Buti M, Colombo M, Pol S, Calinas F, Puoti M, Olveira A, Shiffman M, Stern JO, Kukolj G, Roehrle M, Aslanyan S, Deng Q, Vinisko R, Mensa FJ, Nelson DR. HCVerso1 and 2: faldaprevir with deleobuvir (BI 207127) and ribavirin for treatment-naive patients with chronic hepatitis C virus genotype-1b infection. Clin Exp Gastroenterol. 2016 Nov 24;9:351-363. doi: 10.2147/CEG.S111116. eCollection 2016. PMID 27920566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned that approximately 800 patients would be screened in order to randomize and treat approximately 460 patients (195 patients in treatment Groups 1 and 2 each, 40-70 patients in treatment Group 3).
Pre-assignment Details: Treatment-naïve patients with chronic hepatitis C infection of genotype (GT)1b were included in the trial. Patients with compensated liver cirrhosis, defined as Ishak Grade ≥5 or METAVIR Grade ≥4 on liver biopsy, or liver stiffness of ≥ 13 kilopascal (kPa) on fibroscan, were assigned to Group 3.
Groups:
- 16 wk NC FDV+DBV+RBV: 600 milligram (mg) of Deleobuvir (DBV) twice daily (BID) combined with 240 mg on the first day followed by 120mg of Faldaprevir (FDV) once daily (QD) and 1000-1200mg Ribavirin BID (RBV) for 16 weeks (wk) followed by DBV placebo, FDV placebo and RBV placebo for 8 weeks. All were administered per os (orally).
  This group included non-cirrhotic patients (NC).
- 24 wk NC FDV+DBV+RBV: 600 milligram (mg) of Deleobuvir (DBV) twice daily (BID) combined with 240 mg on the first day followed by 120mg of Faldaprevir (FDV) once daily (QD) and 1000-1200mg Ribavirin (RBV) BID for 24 weeks (wk). All were administered per os (orally).
  This group included non-cirrhotic patients (NC).
- 24 wk CR FDV+DBV+RBV: 600 milligram (mg) of Deleobuvir (DBV) twice daily (BID) combined with 240 mg on the first day followed by 120mg of Faldaprevir (FDV) once daily (QD) and 1000-1200mg Ribavirin (RBV) BID for 24 weeks (wk). All were administered per os (orally). This group comprised patients with compensated cirrhosis (CR) who received open label treatment.
Period: Overall Study
Arm/Group | 16 wk NC FDV+DBV+RBV | 24 wk NC FDV+DBV+RBV | 24 wk CR FDV+DBV+RBV
Started | 208 | 211 | 51
Completed | 162 | 169 | 38
Not Completed | 46 | 42 | 13
Not completed — Adverse Event | 16 | 16 | 4
Not completed — Lack of Efficacy | 21 | 18 | 5
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 8 | 2
Not completed — Other reason not defined above | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The baseline characteristics were carried out on an intent-to-treat basis including all randomized patients who were dispensed study medication and were documented to have taken at least one dose of study medication (FAS).
Groups:
- 16 wk NC FDV+DBV+RBV: 600 mg DBV (BID) + 120mg FDV (QD) + 1000-1200mg RBV (BID) for 16wk followed by DBV placebo, FDV placebo and RBV placebo for 8wk. All were administered per os (orally).
  This group included non-cirrhotic patients (NC).
- 24 wk NC FDV+DBV+RBV: 600 mg DBV (BID) + 120mg FDV (QD) + 1000-1200mg RBV (BID) for 24wk. All were administered per os (orally). This group included non-cirrhotic patients (NC).
- 24 wk CR FDV+DBV+RBV: 600 mg DBV (BID) + 120mg FDV (QD) + 1000-1200mg RBV (BID) for 24wk. All were administered per os (orally). This group comprised patients with compensated cirrhosis (CR) who received open label treatment.
- Total: Total of all reporting groups
Arm/Group | 16 wk NC FDV+DBV+RBV | 24 wk NC FDV+DBV+RBV | 24 wk CR FDV+DBV+RBV | Total
Number analyzed (Participants) | 208 | 211 | 51 | 470
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.1 (12.7) | 51.1 (12.9) | 57.9 (8.8) | 51.4 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 114 | 18 | 254
  Male | 86 | 97 | 33 | 216

OUTCOME MEASURES:

1. Primary Outcome: SVR12 Rates With Historical Control
Description: Sustained Virologic Response at Week 12 post-treatment (SVR12): Plasma Hepatitis C Virus ribonucleic acid (HCV RNA) level <25 international units/millilitre (IU/mL) at 12 weeks after End of Treatment (EoT). SVR12, was assessed based on the observed HCV RNA result taken at least 10 weeks after treatment discontinuation. This definition was also applied to patients who discontinued treatment early: if the patient had HCV RNA undetected at least 10 weeks after stopping all treatment, they were considered a responder in the primary analysis. This is the primary analyses of the primary endpoint
Time Frame: 12 Week (post-treatment)
Population: The primary analyses of efficacy were carried out on an intent-to-treat basis including all randomized patients who were dispensed study medication and were documented to have taken at least one dose of study medication (FAS).
Measure: Number; unit: Percentage of participants
Groups:
- 24 wk FDV+DBV+RBV: 600 mg DBV (BID) + 120mg FDV (QD) + 1000-1200mg RBV (BID) for 24wk (orally) in cirrhotic and non-cirrhotic patients.
- 16 wk FDV+DBV+RBV: 600 mg DBV (BID) + 120mg FDV (QD) + 1000-1200mg RBV (BID), orally. This is the combination of non-cirrhotic patients in the 16 week treatment group and cirrhosis patients in the 24-week treatment group.
Arm/Group | 24 wk FDV+DBV+RBV | 16 wk FDV+DBV+RBV
Number analyzed (Participants) | 262 | 259
Percentage of participants
  non-cirrhotic (N=174, 149) | 82.5 | 71.6
  cirrhotic (N=37, 37) | 72.5 | 72.5
Statistical Analysis 1: Comparison: 24 wk FDV+DBV+RBV; The proportion of patients achieving SVR12 was compared to an acceptable minimum SVR rate achieved with an approved direct acting anti-viral (DAA) in combination with pegylated interferon-alfa (PegIFN) from historical data. The acceptable minimum SVR rate was 71% (reference for PegIFN-eligible); Test type: Superiority or Other; p < 0.0001, Stratified one sample z-test; Adjusted response rate = 81.4, 95% CI 2-sided [76.6 to 86.2] — Adjusted response rate will tested against 71%. It is calculated as a weighted average (non-cirrhotic: 89% times response rate+ cirrhotic: 11% times response rate), 11% is the highest rate of cirrhotic from historical trials with approved DAA+PegIFN
Statistical Analysis 2: Comparison: 16 wk FDV+DBV+RBV; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3989, Stratified one sample z-test; Adjusted response rate = 71.7, 95% CI 2-sided [66.1 to 77.4] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Comparisons of SVR12 Rates Across Treatment Arms
Description: Sustained Virologic Response rates across treatment arms at Week 12 post-treatment (SVR12). This is the secondary analyses of the primary endpoint.
Time Frame: 12 Week (post-treatment)
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | 16 wk NC FDV+DBV+RBV | 24 wk NC FDV+DBV+RBV | 24 wk CR FDV+DBV+RBV
Number analyzed (Participants) | 208 | 211 | 51
Percentage of participants | 71.6 | 82.5 | 72.5
Statistical Analysis 1: Comparison: 16 wk NC FDV+DBV+RBV vs 24 wk NC FDV+DBV+RBV; Test type: Superiority or Other; p = 0.0040, z-test; based on two sample z-test with continuity correction for variance; Koch's method with continuity correction = 10.8, 95% CI 2-sided [2.8 to 18.8]

3. Secondary Outcome: SVR4
Description: Sustained Virologic Response rates across treatment arms at Week 4 post-treatment (SVR4).
Time Frame: 4 Week (post-treatment)
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | 16 wk NC FDV+DBV+RBV | 24 wk NC FDV+DBV+RBV | 24 wk CR FDV+DBV+RBV
Number analyzed (Participants) | 208 | 211 | 51
Percentage of participants
  Percentage of patients with response | 78.4 | 84.4 | 76.5
  Positive predicted value | 94.0 | 98.0 | 95.0
Statistical Analysis 1: Comparison: 16 wk NC FDV+DBV+RBV vs 24 wk NC FDV+DBV+RBV; Category: Percentage of patient with response; Test type: Superiority or Other; p = 0.0575, z-test; based on two sample z-test with continuity correction for variance; Koch's method with continuity correction = 6.0, 95% CI 2-sided [-1.5 to 13.5]

4. Secondary Outcome: SVR24
Description: Sustained Virologic Response rates across treatment arms at Week 24 post-treatment (SVR24).
Time Frame: 24 Week (post-treatment)
Population: FAS
Measure: Number; unit: Percantage of participants
Arm/Group | 16 wk NC FDV+DBV+RBV | 24 wk NC FDV+DBV+RBV | 24 wk CR FDV+DBV+RBV
Number analyzed (Participants) | 208 | 211 | 51
Percantage of participants
  Percentage of patients with response | 70.7 | 80.6 | 72.5
  Positive predicted value | 97.0 | 99.0 | 100.0
Statistical Analysis 1: Comparison: 16 wk NC FDV+DBV+RBV vs 24 wk NC FDV+DBV+RBV; Category: Percentage of patient with response; Test type: Superiority or Other; p = 0.0089, z-test; based on two sample z-test with continuity correction for variance; Koch's method with continuity correction = 9.9, 95% CI 2-sided [1.7 to 18.1]

ADVERSE EVENTS:
Time Frame: From first administration of study medication to 4 weeks after last intake (up to 200 days). Adverse events with an onset date thereafter were to be reported only if serious up to 24 or 48 weeks after last study treatment (up to 340 or 508 days).
Description: Safety analyses were based on the safety set that included all patients who were dispensed study medication and were documented to have taken at least 1 dose of investigational treatment, regardless of randomization.
Arm/Group | 16 wk NC FDV+DBV+RBV | 24 wk NC FDV+DBV+RBV | 24 wk CR FDV+DBV+RBV
Serious Adverse Events (participants affected / at risk) | 7/208 | 11/211 | 4/51
Other Adverse Events (participants affected / at risk) | 192/208 | 198/211 | 49/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 16 wk NC FDV+DBV+RBV (N=208) | 24 wk NC FDV+DBV+RBV (N=211) | 24 wk CR FDV+DBV+RBV (N=51)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0
Gastritis bacterial (Infections and infestations) | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0
Dumping syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Drug abuse (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 16 wk NC FDV+DBV+RBV (N=208) | 24 wk NC FDV+DBV+RBV (N=211) | 24 wk CR FDV+DBV+RBV (N=51)
Anaemia (Blood and lymphatic system disorders) | 40 | 53 | 19
Ocular icterus (Eye disorders) | 20 | 15 | 3
Abdominal discomfort (Gastrointestinal disorders) | 14 | 10 | 3
Abdominal pain (Gastrointestinal disorders) | 14 | 16 | 4
Abdominal pain upper (Gastrointestinal disorders) | 25 | 27 | 2
Constipation (Gastrointestinal disorders) | 12 | 14 | 3
Diarrhoea (Gastrointestinal disorders) | 50 | 66 | 17
Dyspepsia (Gastrointestinal disorders) | 24 | 25 | 5
Nausea (Gastrointestinal disorders) | 96 | 112 | 27
Vomiting (Gastrointestinal disorders) | 64 | 62 | 18
Asthenia (General disorders) | 40 | 58 | 7
Chest pain (General disorders) | 5 | 3 | 3
Chills (General disorders) | 5 | 3 | 3
Fatigue (General disorders) | 53 | 50 | 13
Pyrexia (General disorders) | 6 | 6 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 17 | 17 | 5
Jaundice (Hepatobiliary disorders) | 28 | 35 | 10
Nasopharyngitis (Infections and infestations) | 12 | 13 | 4
Sunburn (Injury, poisoning and procedural complications) | 9 | 17 | 4
Blood bilirubin increased (Investigations) | 8 | 10 | 5
Weight decreased (Investigations) | 13 | 19 | 5
Decreased appetite (Metabolism and nutrition disorders) | 20 | 33 | 6
Vitamin D deficiency (Metabolism and nutrition disorders) | 14 | 21 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 11 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 6 | 1
Dizziness (Nervous system disorders) | 13 | 18 | 5
Dysgeusia (Nervous system disorders) | 11 | 8 | 4
Headache (Nervous system disorders) | 33 | 30 | 4
Paraesthesia (Nervous system disorders) | 11 | 17 | 2
Syncope (Nervous system disorders) | 0 | 8 | 3
Depression (Psychiatric disorders) | 11 | 18 | 1
Insomnia (Psychiatric disorders) | 17 | 29 | 10
Irritability (Psychiatric disorders) | 6 | 14 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 17 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 18 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 9 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 18 | 13 | 2
Erythema (Skin and subcutaneous tissue disorders) | 23 | 28 | 8
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 29 | 30 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 38 | 53 | 20
Rash (Skin and subcutaneous tissue disorders) | 35 | 37 | 11

LIMITATIONS AND CAVEATS:
BI stopped the further development of DBV, per protocol amendment the Follow-up period was reduced to 24 weeks for patients who achieved SVR12, and to 48 weeks for SVR12 non-responders provided they had not started an alternative HCV treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.